CLINICAL TRIAL: NCT03804697
Title: Selective Thromboembolism Prophylaxis After Total Hip Arthroplasty or Total Knee Arthroplasty by a Risk Stratification With Thromboelastography for Asian Populations: A Randomized Control Trial
Brief Title: Selective Thromboembolism Prophylaxis After Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2016-46
Record Dates: First submitted 2018-12-28; First posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2018-12

CONDITIONS: Venous Thrombosis, Deep; Arthroplasty Complications
MeSH Terms: conditions — Venous Thrombosis | interventions — Thrombelastography

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- selective anticoagulation group (Experimental): Selective anticoagulation group used anticoagulant when thromboelastogram（TEG） indicated hypercoagulability.
  TEG was performed 1 day before the surgery, 1 day after the surgery, 3 days after the surgery, and 5 days after the surgery.
  The dosage regimen of anticoagulant was hypodermic injection 0.4 ml low molecular weight heparin per day for 5 days and oral administration of 10 mg Rivaroxaban until one month after the surgery.
  Interventions: Drug: selective anticoagulation
- conventional anticoagulation group (Active Comparator): The Intervention for conventional anticoagulation group was using anticoagulant until one month after surgery routinely.
  The dosage regimen of anticoagulant was hypodermic injection 0.4 ml low molecular weight heparin per day for 5 days and oral administration of 10 mg Rivaroxaban until one month after the surgery.
  Interventions: Drug: selective anticoagulation

INTERVENTIONS:
Drug: selective anticoagulation — Selective anticoagulation group used anticoagulant once thromboelastography indicated hypercoagulable state. Conventional anticoagulation group used anticoagulant until one month after surgery routinely. The main difference was that the experimental group did not use anticoagulation if the thromboelastography indicated that the blood coagulation status was normal while the control group use anticoagulation routinely.
  Other Names: Thromboelastography

SUMMARY:
Asian populations have a lower rate of high-risk gene mutations of venous thrombosis, which means a reasonable perioperative anticoagulant management after hip or knee arthroplasty for Caucasian populations may be too excessive for Asians. So, individual patient risk assessment, rather than a "blanket policy", is considered the best thromboembolism prophylaxis for Asians.The purpose of this study was to evaluate the effectiveness and safety of selective thromboembolism prophylaxis compared with conventional thromboembolism prophylaxis by risk stratification with thromboelastography (TEG) after joint arthroplasty for Asian populations.

DETAILED DESCRIPTION:
Asian patients who underwent hip or knee arthroplasty in Guangdong General Hospital from August 2016 to August 2017 were randomly divided into selective anticoagulation group (SAG) and conventional anticoagulation group (CAG). SAG used anticoagulant when TEG indicated hypercoagulability while CAP used anticoagulant until one month after surgery regularly. Data including patients' basic information, postoperative complications, perioperative clotting index, intraoperative blood loss, perioperative TEG, volume of drainage, and blood transfusion were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age,
* ASA Ⅰ-Ⅱ grade,
* BMI <40Kg / M ^ 2
* Underwent total knee arthroplasty/ total hip arthroplasty in Guangdong General Hospital
* consent to enroll in this study

Exclusion Criteria:

* history of VTE, preoperative infection, preoperative coagulation
* liver and kidney function existed clinically abnormalities
* history of tumor
* history of vascular surgery
* heart infarction or cerebral infarction within 6 months
* history of lower extremity surgery within 3 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
The Incidence of Deep Vein Thrombosis | 1 day after surgery
  Measured by ultrasound,
The Incidence of Deep Vein Thrombosis | 3 days after surgery
  Measured by ultrasound
The Incidence of Deep Vein Thrombosis | 5 days after surgery
  Measured by ultrasound
The Incidence of Deep Vein Thrombosis | 1 month after surgery
  Measured by ultrasound
The Incidence of Deep Vein Thrombosis | 3 months after surgery
  Measured by ultrasound
The Incidence of Deep Vein Thrombosis | 6 months after surgery
  Measured by ultrasound

SECONDARY OUTCOMES:
Hematocrit | 1 day before surgery
  Measured by Complete Blood Count
Hematocrit | 1 day after surgery
  Measured by Complete Blood Count
Hematocrit | 3 days after surgery
  Measured by Complete Blood Count
Hematocrit | 5 days after surgery
  Measured by Complete Blood Count
Hemoglobin | 1 day before surgery
  Number of Hemoglobin Measured by Blood Test
Hemoglobin | 1 day after surgery
  Number of Hemoglobin Measured by Blood Test
Hemoglobin | 3 days after surgery
  Number of Hemoglobin Measured by Blood Test
Hemoglobin | 5 days after surgery
  Number of Hemoglobin Measured by Blood Test
Red Blood Cell | 1 day before surgery
  Number of Red Blood Cell Measured by Complete Blood Count
Red Blood Cell | 1 day after surgery
  Number of Red Blood Cell Measured by Complete Blood Count
Red Blood Cell | 3 days after surgery
  Number of Red Blood Cell Measured by Complete Blood Count
Red Blood Cell | 5 days after surgery
  Number of Red Blood Cell Measured by Complete Blood Count
Volume of Transfusion | During Hospitalization
  Volume of Blood Transfusion
Transfusion Rate | During Hospitalization
  Number of patients who receive transfusion divided by total number of patients in the group
Superficial Infection | During Hospitalization
  Number of patients who suffer superficial infection
Superficial Infection | 1 month after surgery
  Number of patients who suffer superficial infection
Superficial Infection | 3 months after surgery
  Number of patients who suffer superficial infection
Superficial Infection | 6 months after surgery
  Number of patients who suffer superficial infection
Deep Infection | During Hospitalization
  Number of patients who suffer deep infection
Deep Infection | 1 month after surgery
  Number of patients who suffer deep infection
Deep Infection | 3 months after surgery
  Number of patients who suffer deep infection
Deep Infection | 6 months after surgery
  Number of patients who suffer deep infection
Ecchymosis incidence Rate | 1 month after surgery
  Number of patients who suffer ecchymosis divided by total number of patients in the group